CLINICAL TRIAL: NCT05709262
Title: Comparison of Different Walk and Performance Test in Detecting Silent Hypoxia in SARS-CoV-2
Brief Title: Comparison of Different Walk and Performance Test in Detecting Silent Hypoxia
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Ismail Saracoglu, Director, Kutahya Health Sciences University
Other Study IDs: KSBUSilentHypoxi
Record Dates: First submitted 2023-01-03; First posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Hypoxia; COVID-19 Pneumonia; Oxygen Saturation; Pulmonary Rehabilitation
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Healthcare systems around the world have been dealing with COVID 19. One of the main manifestations of this infection is lung involvement of varying degrees, causing a spectrum of diseases from mild lower respiratory tract infection to severe Adult Respiratory Distress Syndrome (ARDS). One of the important clinical parameters is to detect hypoxia early in order to initiate a higher level of care at the earliest. The presence of silent or latent hypoxia has made this task difficult in COVID 19. Besides, critical findings such as silent hypoxia that is not at rest but triggered by effort can be revealed by some practical field tests such as the 6-minute walk test or the 1-minute chair sit and stand test. Moreover, these simple tools also help to investigate the patient's readiness for discharge. In this way, it will be useful to evaluate their usability in discharge decisions or in determining the post-discharge cardiopulmonary reserves of the patients and therefore their rehabilitation needs. Although walk and performance tests can be performed naturally, safely and simply, more similarly to movements in daily living activities compared to cardiopulmonary exercise tests, the interest in these tests has increased over the years, especially in subjects such as exercise capacity, mortality and morbidity expectation, or oxygen desaturation in patients with chronic cardiopulmonary pathology. The number of studies in 19 patients is quite limited. For this reason, the necessity of new studies on different field tests to detect the presence of latent hypoxia, which expresses the oxygen desaturation triggered by effort, and to evaluate the exercise tolerance status before discharge, has been emphasized in recent reviews.The aim of this study is to determine the presence of silent hypoxia, which expresses the oxygen desaturation triggered by effort, in Covid-19 patients and to compare the different short-term walk and performance tests, which the investigators consider easier and applicable in the conditions of the pandemic environment, with the classical gold standard test ( Six minute walk test) in order to evaluate the exercise tolerance status of the patients before discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of covid 19 between the ages of 18-80
* Patients with a SaO2 value > 93 in room air
* Patients who do not have dyspnea symptoms in room air during rest
* Patients whose breathing frequence < 21 at rest
* Patients who can walk independently and get up from their seat
* Patients who did not receive any rehabilitation
* Patients who can cooperate and who are fully oriented
* Patients who volunteered to participate in the study

Exclusion Criteria:

* Severe pnemonia due to Covid-19
* Exacerbation, severe respiratory failure (resting partial pressure of oxygen in standard ambient conditions of less than 55 mmHg), and inability or unwillingness to understand or comply with the study protocol.
* Unable to walk unaided
* Patients diagnosed with vertigo, Meniere, etc. balance disorder and dizziness
* Patients diagnosed with orthostatic hypotension
* Patients diagnosed with neurologic disease such as: stroke, ms-like neuromotor pathology
* pregnant women and those diagnosed with epilepsy
* Patients with BMI > 35
* Patients with problems in cooperation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will consist of Covid-19 patients hospitalized in the pandemic wards of Kütahya Health Sciences University Physical Medicine and Rehabilitation Additional Service building.
  All volunteer patients who meet our inclusion and exclusion criteria will undergo walking field tests with at least 2 hours between them after their written consent is obtained.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-12-19 (Actual); Primary Completion 2022-04-19 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
Six minute walk test | 10 minutes
  The six-minute walk test is a submaximal exercise test that can be safely performed even by patients with heart failure who cannot tolerate the maximal exercise test. The test is very simple, requires inexpensive equipment, and is reproducible. In addition, it is considered safe as patients are self-limiting during exercise. The 6-minute walk test, which is performed in diseases such as pulmonary hypertension and COPD, is simply used to show the shortness of breath on exertion and the exercise capacity of the patient. In the 6-minute walking test, the patient is preferably walked along a straight corridor of at least 30 meters as fast as he can, but without running. Measure how many meters patients walk.
Two minute walk test | Baseline
  The Two Minute Walk Test is a measure of self-paced walking ability and functional capacity, particularly for those who cannot manage the longer Six Minute Walk Test.
Fourty step walk test | Baseline
  Patients are asked to take 40 steps and time is kept. At the same time, oxygen desaturations are checked. This test, which is widely used in the triage and discharge evaluation of Covid-19 patients, especially in the UK, and aims to detect exertional desaturation, has not been validated in any disease yet, but it can be applied even at home in current reviews because it requires less effort and is found to be quite safe compared to other tests. highlighted as a test. On the other hand, the sensitivity was expressed as low because it was not a compelling test.
30 Second Sit to Stand Test | Baseline
  The 30 Second Sit to Stand Test is also known as 30 second chair stand test, is for testing endurance. It is part of the Fullerton Functional Fitness Test Battery. To determine the oxygen saturation, the patient is observed with the pulse saturation probe for 1 minute after the test.
1 Minute Sit to Stand Test | Baseline
  The 1-min sit-to-stand test evaluate in mild COVID-19 cases (not requiring intensive care unit admission on initial evaluation if their SpO2 was more than 95% while breathing ambient air.

SECONDARY OUTCOMES:
Vital measurements before, during and after walk test | Baseline
  Patients will wear a mobile pulse oximeter that continuously recorded heart rate and oxygen saturation. The device will used to record breathing frequency via a nasal cannula. Baseline values of oxygen saturation, heart rate, breathing frequency, and ratings of perceived exertion on the modified Borg scale (0-10) for dyspnea and leg fatigue will be recorded before, during and immediate after walk tests.

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Saracoglu, Principal Investigator — Kutahya Health Sciences University
Locations (1):
- Kutahya Health Sciences University Evliya Celebi Hospital Physical Therapy and Rehabilitation Department, Kütahya, Turkey (Türkiye)